CLINICAL TRIAL: NCT00522431
Title: An Open Label Phase 3 Study of Fortigel Testosterone Gel 2% in Hypogonadal Males
Brief Title: A Study of Fortigel Testosterone Gel 2% in Males With Low Testosterone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOR01C
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Hypogonadism
Keywords: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

ARMS (1):
- 1 (Experimental): 2% testosterone gel
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — 2% gel
  Other Names: Fortigel

SUMMARY:
Low testosterone is a condition that occurs when the body is unable to produce sufficient quantities of testosterone. The medical name for low testosterone is hypogonadism. Hypogonadism can be caused by many factors. Symptoms include: decrease in libido, lack of energy and mood swings. The goal of testosterone replacement therapy is to return testosterone levels to the normal range and relieve symptoms.

The purpose of this study is to evaluate the ability of Fortigel testosterone gel 2% to maintain serum (blood) testosterone levels within the normal range in hypogonadal men aged 18 to 75 years. This will be determined by blood sampling at specified times during the study. The study is also intended to evaluate the tolerability of Fortigel, which will be applied to the skin each day throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 - 75 years with primary or secondary hypogonadism as confirmed by:

  * Single serum total testosterone concentration < 250 ng/dL, or
  * Two consecutive serum total testosterone concentrations < 300 ng/dL (determined at least one week apart during the screening period).
* Has a BMI ≥ 22 kg/m2 and < 35 kg/m2.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2007-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liz Waldie, Study Director — Strakan Pharmaceuticals, Inc.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 406 participants screened, 149 met the inclusion/exclusion criteria and entered the study.
Groups:
- Fortigel: 40 mg testosterone in 2 g gel applied topically once daily for 90 days (adjusted to between 10 and 70 mg per day)
Period: Overall Study
Arm/Group | Fortigel
Started | 149
Completed | 138
Not Completed | 11
Not completed — Adverse Event | 5
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 2
Not completed — Subject non-compliance | 1
Not completed — Other/unknown | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Fortigel
Number analyzed (Participants) | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 149

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Meeting Serum Total Testosterone Average Concentration (Cavg) Criteria at Day 90
Description: Percentage of participants with Cavg0-24h ≥300-≤1140 ng/dL
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 10, 12 and 24 hours after study drug application on day 90
Population: Modified intent-to-treat (mITT) population included participants who had more than 1 pharmacokinetic (PK) sample obtained during the 24-hour PK profile on day 90 (11 participants were excluded); data from 9 additional participants were excluded due to insufficient backup samples needed for reanalysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fortigel
Number analyzed (Participants) | 129
percentage of participants | 77.5 [70.3 to 94.7]

2. Secondary Outcome: Percentage of Participants Meeting Serum Total Testosterone Maximum Concentration (Cmax) Criteria at Day 90
Description: Percentage of participants with Cmax ≤1500 ng/dL, 1800-2500 ng/dL, and >2500 ng/dL
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 10, 12 and 24 hours after study drug application on day 90
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Fortigel
Number analyzed (Participants) | 129
percentage of participants
  ≤1500 ng/dL | 94.6
  1800-2500 ng/dL | 1.6
  >2500 ng/dL | 0

ADVERSE EVENTS:
Time Frame: Throughout the study (approximately 93 days)
Arm/Group | Fortigel
Serious Adverse Events (participants affected / at risk) | 5/149
Other Adverse Events (participants affected / at risk) | 67/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fortigel (N=149)
Intestinal obstruction (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fortigel (N=149)
Skin reaction (Skin and subcutaneous tissue disorders) | 25
Rash (Skin and subcutaneous tissue disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 10
Sinusitis (Infections and infestations) | 6
Cellulitis (Infections and infestations) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Haematuria (Renal and urinary disorders) | 2
Prostatic specific antigen increased (Investigations) | 2
Hypertension (Vascular disorders) | 4
Abnormal dreams (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication statement in clinical trial agreement